CLINICAL TRIAL: NCT02368522
Title: Comparative Assessment of Utilization of Antiviral Therapies in Hepatitis C and Effectiveness of Daclatasvir-containing Regimens in Real-life Clinical Care in Europe
Brief Title: Comparative Assessment of Utilization of Antiviral Therapies in Hepatitis C and Effectiveness of Daclatasvir-containing Regimens in Real-life Clinical Care in Europe (CMPASS-EU)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-259
Record Dates: First submitted 2015-02-12; First posted 2015-02-23 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with and without exposure

SUMMARY:
The study aims to collect information on the current treatment patterns for Hepatitis C in participating countries. There is also a focus on patients receiving a daclatasvir-containing treatment regimen who will be followed prospectively for 12 months after treatment initiation to collect real-world data on effectiveness and safety of the treatment. Additional analysis will differentiate between selected subpopulations.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Adult (≥18 years at inclusion)
* Diagnosed with a chronic hepatitis C infection
* Whose physician has already decided to initiate a new HCV treatment or a new daclatasvir-containing regimen
* Informed consent to participate in the study

Exclusion Criteria:

* Participation in a clinical trial or an early access program for HCV therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from private practices and outpatients units in hospitals
Sampling Method: Probability Sample
Enrollment: 920 (Actual)
Dates: Start 2014-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Quantify effectiveness of daclatasvir (DCV) containing regimen overall and in subgroups (GT1, non GT1 and cirrhotic patients) by measuring sustained virologic response (SVR12) | Upto week 12 after the end of HCV treatment (SVR12)
  SVR12 defined as a documented undetectable viral load on or after week 12 following the end of treatment

SECONDARY OUTCOMES:
SVR12 in patients treated with DCV-containing regimens in real-life by treatment regimen, genotype, cirrhosis stage, HCV-treatment experience, HIV coinfection, and previous LTx (if present) | Upto week 12 after the end of HCV treatment (SVR12)
Proportion of patients on DCV-containing regimens achieving SVR12 in real-life compared with SVR12 rates in clinical trials | Upto week 12 after the end of HCV treatment (SVR12)
Safety of DCV-containing regimens in real-life measured by the incidence of (S)AEs and the incidence leading to treatment discontinuation | Until completion of study
Demographic and clinical characteristics and treatment patterns of patients starting a new HCV treatment regimen (with or without DCV), overall and by treatment regimen,GT,cirrhosis stage,HCV-treatment experience,HIV co-infection,and previous LTx | Baseline (single assessment)
  Previous LTx (if present)
Comparison of demographic and clinical characteristics of patients starting a new HCV treatment regimen (with or without DCV) by treatment regimen and to identify factors associated with the initiation of different regimens | Baseline (single assessment)
SVR 24 in patients treated with DCV-containing regimens in real-life clinical care, change of Child-Pugh Score and Metavir score as well as change of patient related outcomes (EQ-5D and SF-36 questionnaires measuring quality of life) | Upto week 24 after the end of HCV treatment (SVR24)
  Metavir score (liver function and histology)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hamburg, Germany

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx